CLINICAL TRIAL: NCT06639464
Title: Semaglutide for the Treatment of Opioid Use Disorder: A Pilot Randomized Controlled Trial
Brief Title: Semaglutide for Helping Opioid Recovery
Acronym: SHORE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Director, Division of Addiction Psychiatry, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024P002669
Record Dates: First submitted 2024-09-20; First posted 2024-10-15 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder
Keywords: semaglutide; opioid use disorder; buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The IDS will perform both the randomization and blinding, and will be the only research staff that will remain unblinded. The IDS will extract the semaglutide and draw the dose into syringes, which will be made to match visually with the placebo saline doses. All other research staff will remain blinded for the duration of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental): This arm will receive semaglutide (n=23). All participants will initially receive 0.25mg for 4 weeks, and then as tolerated dose will be increased to 0.5mg for 4 weeks. Then as tolerated, the dose will be increased to 1.0mg for 4 weeks.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): This arm will receive saline placebo (n=23).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Semaglutide — This intervention will consist of the FDA-approved dosing schedule, with terminal dosage based on manufacturer's recommendation to titrate to 1mg over 12 weeks. Participants will receive 0.25mg for the first 4 weeks, 0.5mg for the next 4 weeks, and 1.0mg for the final 4 weeks. IDS will extract semaglutide an draw the doses into syringes for matching placebo doses to also be produced and maintain blind.
  Other Names: Ozempic
  Arms: Semaglutide
Other: Placebo — Placebo syringes of saline and matching volume will be produced by IDS.
  Arms: Placebo

SUMMARY:
The is a pilot, 12-week, double-blind, placebo-controlled, randomized trial of individuals with opioid use disorder (OUD) newly initiating buprenorphine to receive either weekly injections of semaglutide (n=23) or matching placebo (n=23). The primary aim is to determine the effects of semaglutide on cue-reactivity among individuals with OUD. The secondary aim is to assess the preliminary efficacy, safety, and tolerability of semaglutide for OUD.

DETAILED DESCRIPTION:
Participants include N=46 men and women with DSM5 diagnosis of OUD who are newly initiating sublingual buprenorphine (SL-BUP), defined as within 60 days of enrollment. Only those participants who have attained stable SL-BUP dosing (i.e. no change in dose) for at least 30 days prior to enrollment and plan to remain on the SL-BUP for the duration of the trial will be eligible. Potential participants will be screened and enrolled only if they meet full inclusion criteria. After baseline procedures are complete, participants will be randomized to semaglutide or placebo. Following randomization, participants will be scheduled for thirteen weekly study visits. Each visit will last approximately 1 hour, except for study visits 1 (baseline), 7, and 14 (follow-up) which will take no more than 3 hours in order to conduct reward- and stress-related neurocognitive testing. At each visit, participants will complete vital signs, weight, urine toxicology testing, and a blood testing for glucose. Participants will also complete an assessment of adverse events and questionnaires probing secondary outcomes (i.e. anxiety and depression, suicidality, substance use, opioid withdrawal symptoms, craving questionnaire). Blood samples will be collected at the beginning, middle, and end of the study. At study visits 2-13, the weekly dose of semaglutide or placebo will be administered. Both participants and study staff (including raters) will be blinded to active drug vs. placebo. The medication will be purchased from the manufacturer, and stored in the BWH Investigational Drug Service (IDS). The IDS will then extract the semaglutide and draw the dose into syringes, which will be matching visually with the placebo doses.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults aged 18 and above
* DSM-5 diagnosis of opioid use disorder, severe
* Initiated sublingual buprenorphine (SL-BUP) treatment within 60 days of enrollment
* Attained stable dosing of SL-BUP of 16mg or greater for 30 days prior to enrollment
* Anticipating continuation of SL-BUP for the duration of the trial
* Agreeable with bringing SL-BUP prescription to visits to allow study team to conduct a dose count
* Willing to grant study team permission to communicate about SL-BUP treatment with community prescriber via completion of 42 CFR release

Individuals with any of the following will be excluded:

* DSM-5 diagnosis of any current substance use disorder excluding opioid, cannabis or tobacco
* Active psychosis, active suicidality or homicidality or any psychiatric condition that impair ability to provide informed consent
* Any current or lifetime diagnosis of eating disorders
* BMI<25mg/kg2
* Current or lifetime diagnosis of Type 1 or Type 2 diabetes
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
* Use of any GLP-1 agonist medications in the prior 3 months
* Anticipating receipt of any GLP-1 agonist medications during the trial
* History of angina pectoris, coronary heart disease, congestive heart failure, inflammatory bowel disease, chronic obstructive pulmonary disease, bariatric surgery, idiopathic pancreatitis, diabetic gastroparesis
* Liver function test greater than 3 times upper normal limit
* Renal impairment as indicated by eGFR of <60
* History of hypersensitivity or allergy to semaglutide
* Pregnant or breastfeeding
* Anticipated to participate in a concurrent drug trial
* Any other reason or clinical condition that the investigators judge may interfere with study participation and/or be unsafe for a participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Cue-induced Cravings for Opioids | Baseline, 6 weeks, and 13 weeks after baseline visit
  Cue-induced craving scores at study completion compared to baseline using a standard cue-reactivity paradigm utilizing visual cues. Cravings will be measured on a scale from 0-10 with 10 meaning extreme cravings.
Relapse to Illicit Opioid Use | Weekly from baseline to end of study at 14 weeks
  the primary outcome is proportion of participants who relapse to illicit opioids use at study completion, defined as the start of 4 consecutive opioid "use weeks" or at the start of 7 consecutive days of self-reported opioid use days. A "use week" is defined as any week in which participants self-report at least one day of illicit opioid use, provide a urine test positive for illicit opioids, or fail to provide a urine sample for testing. The study investigators will use Time-Line Follow Back (TLFB), a gold-standard method of evaluating substance use, as well as weekly urine toxicology screens.

SECONDARY OUTCOMES:
Visual Probe Task | Baseline, 6 weeks, and 13 weeks after baseline visit
  A behavioral task to assess attentional bias. Opioid-related and neutral images will be used, different from the ones used for the cue-reactivity paradigm to limit habituation. A pair of images will appear on the left and right of the screen for either a short (200ms) or long (500ms) stimulus duration to assess automatic orientating and controlled attention processing, respectively. Image pairs will be replaced by a probe in the location of either the opioid-related or neutral image. The probe will remain until the participant responds to identify the probe orientation by pressing the response keys as quickly as possible. This task will yield reaction times for analysis.
Iowa Gambling Task (IGT) | Baseline, 6 weeks, and 13 weeks after baseline visit
  A computerized task to measure risky decision making using four decks of cards (A, B, C, D). Participants are instructed to maximize profits. Cards from decks A and B earn more profits but lead to even higher occasional losses leading to net long-term losses, while decks C and D yield low profits but only low occasional losses resulting in a net long-term profit. The task will yield scores which are the sums of cards selected from decks A/B and decks C/D.
Monetary Choice Questionnaire (MCQ) | Baseline, 6 weeks, and 13 weeks after baseline visit
  A self-report tool used to measure delayed discounting. Participants will be asked to pick one of the two choices given. Score calculated typically falls between 0.0 and 0.5, with smaller values indicating a lack of discounting and preference for delayed rewards and higher values indicating strong discounting and a preference for immediate rewards.
Clinical Opiate Withdrawal Scale (COWS) | Weekly from baseline to end of study at 14 weeks
  Tool for assessing opioid withdrawal. Scale of 0-48, with a higher number meaning more severe withdrawal.
Patient Health Questionnaire (PHQ8) | Weekly from baseline to end of study at 14 weeks
  A tool to assess depression symptoms. Scale of 0-24, with a higher score meaning more depression symptoms.
Generalized Anxiety Disorder (GAD7) | Weekly from baseline to end of study at 14 weeks
  A standard tool to assess anxiety symptoms. Scale of 0-21 with a higher number indicating more anxiety.
WHO Quality of Life (WHOQOL-BREF) | Baseline and 13 weeks after baseline visit
  A 26-item quality of life scale. Split into 5 domain scores: Overall Quality of Life and General Health (2-10), Physical Health (7-35), Psychological (6-30), Social relationships (3-15), and Environment (8-40). Higher scores indicate a higher quality of life.
Patient Rated Inventory of Side Effects (PRISE) | Weekly from 2 weeks after baseline to end of study at 14 weeks
  A self-report tool to qualify side effects. For each domain, the patient rates whether the symptoms are tolerable or distressing.
Hemoglobin A1c | At baseline and 13 weeks after baseline visit
  Hemoglobin A1c levels will be obtained via blood draw
Stanford Efficacy of treatment Scale (SETS) | Baseline
  An instrument for measuring patient outcome expectancy in clinical trials. Assesses positive and negative treatment expectations with 3 items each on 7-point Likert-scales from 0 'not agree at all' to 6 'fully agree'.
Columbia suicide severity rating scale (C-SSRS) | Weekly from baseline to end of study at 14 weeks
  A commonly used tool to assess suicidal ideation. The sum ranges from 2 to 25, with the higher number indicating more intense ideation.
Heart Rate | Weekly from baseline to end of study at 14 weeks
  Heart rate measured in beats per minute (bpm).
Opioid Craving Scale | Weekly from baseline to end of study at 14 weeks
  3-item measure of craving for opioids. Each item will be measured on a scale from 0-10 with 10 meaning stronger cravings.
Blood pressure | Weekly from baseline to end of study at 14 weeks
  Blood pressure measured as (systolic)/(diastolic).
Blood sugar | Weekly from baseline to end of study at 14 weeks
  Blood glucose
Assessment of blind | 6 weeks and 13 weeks after baseline visit.
  Measure of participant perception of whether they received the active study drug.
Height | Weekly from baseline to end of study at 14 weeks
  Height measured in meters.
Weight | Weekly from baseline to end of study at 14 weeks
  Weight measured in kilograms.
Temporal Experience of Pleasure Scale (TEPS) | At baseline and 13 weeks after baseline visit
  A tool to assess both anticipatory and consummatory reward. 18-item tool where each item is ranked from 1 ('very false for me') to 6 ('very true for me'). Items are averaged, with higher score indicate a stronger tendency to anticipate or experience pleasure.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided